CLINICAL TRIAL: NCT05027412
Title: Transurethral En Bloc Resection With Collins Loop vs Conventional Transurethral Resection for the Treatment of Urothelial Bladder Carcinoma
Brief Title: En Bloc TURBT With Collins Loop vs Conventional TURBT
Acronym: TURBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Fuenlabrada (Other)
Responsible Party: Principal Investigator, Berta Nasarre, Attending Physician, Hospital Universitario de Fuenlabrada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URO
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer; Bladder Neoplasm; Bladder Urothelial Carcinoma; Bladder Cancer Stage; Urothelial Carcinoma Recurrent
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- En Bloc TURBT with Collins Loop (Experimental): If the patient is randomized to the TURB group, it will be carried out with a Collins loop, with bipolar energy.
  After randomization, demographic data (age, sex, exposure to tobacco, occupational risk), symptoms prior to randomization (micro or macrohematuria, LUTS) and laboratory data (urinary cytology, hemoglobin and serum creatinine) will be collected. Finally, the physical characteristics of the lesion will be noted in the cystoscopy immediately prior to the intervention: size, location (s) and appearance of the tumor. After the intervention, the type of procedure (TURB / TUB), the duration of the procedure from when the resector is inserted until the urinary catheter is placed, and complications according to the Clavien-Dindo scale will be recorded. In your first post-surgical check-up, the days of hospital stay and the time of bladder catheterization will be collected.
  Interventions: Device: En bloc TURBT Collins Loop
- Conventional TURBT (Active Comparator): The TURB will be carried out with bipolar current according to the traditional technique.
  Interventions: Device: Conventional TURBT

INTERVENTIONS:
Device: En bloc TURBT Collins Loop — En bloc TURBT Collins Loop
  Arms: En Bloc TURBT with Collins Loop
Device: Conventional TURBT — Conventional TURBT
  Arms: Conventional TURBT

SUMMARY:
This is a prospective, randomized, randomized and single-blind study in patients diagnosed with primary bladder CV. Patients diagnosed by cystoscopy of a bladder tumor and with indication for endoscopic surgical treatment, who meet the inclusion criteria, and who sign the Informed Consent (IC), will be randomized.

DETAILED DESCRIPTION:
The main objective of the study is to assess the quality of the resection, defined as the presence of detrusor muscle in the resected tissue.

The secondary objetives are:

* Compare the surgical time, hospital stay, urinary catheterization time and incidence of complications.
* Compare tumor recurrence after one year of follow up.
* Determine the number of re-TURB as a consequence of the absence of muscle layer in the sample or artifacts (Tx)
* Establish the incidence of conversions as a consequence of difficulties in the technique or intraoperative bleeding.
* Compare the degree of satisfaction of the surgeon

ELIGIBILITY:
Inclusion Criteria:

* >18 years old.
* Polypoid / sessile primary tumor.
* < 3 tumors
* Tumor size 10 - 30 mm.

Exclusion Criteria:

* > 4 tumors
* Size of the largest tumor <1 cm and> 4 cm.
* Tumor located in the bladder dome.
* No visualization of the ureteral meatus.
* Flat or in situ tumor.
* Non-urothelial tumors.
* Clotting disorder or treatment with oral anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
presence of detrusor muscle in the resected sample | 1 year of follow up
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: emilio f ripalda, MD, Principal Investigator — Hospital Universitario de Fuenlabrada
Locations (1):
- Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No